CLINICAL TRIAL: NCT01404845
Title: Assessment of the Evolution of Macular Pigment Density in Two Distinct Populations, Before and After Supplementation With Nutrof Total Versus Dietary Supplement Without Lutein and Zeaxanthin, Using the Macular Pigment Module of Visucam 200 or Visucam 500 (Zeiss).
Brief Title: Macular Pigment Density Evolution in Unilateral Wet AMD Versus Non AMD Patients With or Without Lutein and Zeaxanthine Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affordance (Network)
Collaborators: Drescode (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2011-A00922-39
Record Dates: First submitted 2011-07-22; First posted 2011-07-28 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: exudative AMD; dietary supplements; macular pigment; lutein; zeaxanthin; Nutrof total; in one eye
MeSH Terms: interventions — Dietary Supplements; Lutein; Zeaxanthins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B: patients with wet AMD in one eye. (Active Comparator): group B: patients with wet AMD in one eye. In each group, A and B, half the patients will be randomized in a subgroup to Nutrof Total, and the other half in a subgroup to a food supplement not containing Lutein and Zeaxanthin.
  Interventions: Dietary Supplement: Nutrof Total; Dietary Supplement: food supplement without Lutein and Zeaxanthin
- A :patients without retinal pathology (Active Comparator): group A :patients without retinal pathology who underwent cataract surgery 1 month previously.
  In each group, A and B, half the patients will be randomized in a subgroup to Nutrof Total, and the other half in a subgroup to a food supplement not containing Lutein and Zeaxanthin.
  Interventions: Dietary Supplement: Nutrof Total; Dietary Supplement: food supplement without Lutein and Zeaxanthin

INTERVENTIONS:
Dietary Supplement: Nutrof Total — Nutrof Total : 2 capsules per day,during 8 months (5 mg Lutéine + 1 mg Zéaxanthine / capsule).
Dietary Supplement: food supplement without Lutein and Zeaxanthin — food supplement without Lutein and Zeaxanthin : 2 capsules per day, during 8 months.

SUMMARY:
•Purpose: Age-related Macular Degeneration ( AMD) is the leading cause of blindness and visual impairment in industrialized countries. The macular pigment, composed of carotenoid derivatives (lutein and zeaxanthin), may play an important role in the occurrence of AMD. An increase in macular pigment following dietary supplementation with lutein and zeaxanthin could allow early treatment with such supplements in subjects with a high risk of AMD, and encourage them to change their eating habits.

•Primary outcome:

Comparative analysis of the density and evolution of the density of macular pigment:

* In patients without any retinal pathology who underwent cataract surgery 1 month previously
* In the non-exudative eye of patients with exudative AMD in one eye by analyzing the density and evolution of the density of macular pigment in the non-exudative eye

  * Secondary outcomes:

Analysis of changes in macular pigment density after taking food supplements (Nutrof Total versus comparator):

* Time taken to reach the maximum plateau of macular pigment density (no increase in density between 2 measurements)
* Time taken to return to the baseline macular pigment density after cessation of supplementation

  * Study design :

Pilot study -Prospective, randomised, double-masked, comparative, multicenter.

ELIGIBILITY:
Inclusion criteria:

* Both genders (male or female), ≥ 55 years of age.
* Patients without any retinal pathology who underwent cataract surgery 1 month previously Or
* Patients with neovascular AMD (Age-related macular Degeneration) in one eye.
* Patients who gave their written consent

Exclusion Criteria:

Exclusion criteria related to the study:

* Intolerance to the tested product
* Change in fundus image
* Patients already taking Nutrof Total or similar supplements containing Lutein and Zeaxanthin
* Allergy to mydriatics

Exclusion criteria for ophthalmologic reasons:

o Ocular diseases or conditions whose presence might interfere with the measurement of optical density of macular pigment (e.g. cataract, diabetic retinopathy, optic atrophy, myopia> -6.5 Diopters)

Exclusion criteria for systemic reasons:

o Medical or surgical history, disorder or disease (e.g. severe organic disease, acute or chronic: liver disease, endocrine, neoplastic, hematologic, infectious diseases, severe psychiatric disorder, significant cardiovascular abnormalities, etc...) and / or aggravating factors or structural defect, considered as being inconsistent with the study by the investigator.

Exclusion criteria for general reasons:

* Inability of the patient to understand the study procedures and to give informed consent.
* Ward of court
* Patient not covered by the social security scheme
* Pregnancy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Comparative analysis of macular pigment density | 18 months
  Comparative analysis of macular pigment density in patients who underwent cataract operation 1 month ago, without retinal pathology and in patients with exudative AMD in one eye by analyzing the density and evolution of the density of macular pigment in the non-exudative eye.
  Optical density (OD)parameters of the macular pigments measured by an objective reflectometry method based on a 30° field image acquired by the Visucam 200 or 500 of Zeiss :
  Area : where macular pigments could be detected
  Max OD/Mean OD/ Volume : Maximum value/Mean Value/Sum of all OD in the area

SECONDARY OUTCOMES:
Analysis of changes in macular pigment density | 18 months
  Analysis of changes in macular pigment density after taking food supplements (Nutrof Total versus comparator):
  * Time taken to reach the maximum plateau of macular pigment density (no increase in density between 2 measurements)
  * Time taken to return to the baseline macular pigment density after cessation of supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Martine Mauget-faysse, Principal Investigator — Affordance
Locations (2):
- France (2):
  - Docteur Jean-Jacques Masella, Grenoble
  - Centre ophtalmologique Rabelais, Lyon

REFERENCES:
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Delcourt C. Epidémiologie de la DMLA dans la population française. In: Soubrane G, Coscas G, Souied EH, editors. Les DMLAs (9ème édition). Rapport de la Société Française d'Ophtalmologie. Paris: Masson; 2007. p. 108-110.
- [Background] Jager RD, Mieler WF, Miller JW. Age-related macular degeneration. N Engl J Med. 2008 Jun 12;358(24):2606-17. doi: 10.1056/NEJMra0801537. No abstract available. PMID 18550876
- [Background] Age-Related Eye Disease Study Research Group. A randomized, placebo-controlled, clinical trial of high-dose supplementation with vitamins C and E, beta carotene, and zinc for age-related macular degeneration and vision loss: AREDS report no. 8. Arch Ophthalmol. 2001 Oct;119(10):1417-36. doi: 10.1001/archopht.119.10.1417. PMID 11594942
- [Background] Whitehead AJ, Mares JA, Danis RP. Macular pigment: a review of current knowledge. Arch Ophthalmol. 2006 Jul;124(7):1038-45. doi: 10.1001/archopht.124.7.1038. PMID 16832030
- [Background] Antioxidant status and neovascular age-related macular degeneration. Eye Disease Case-Control Study Group. Arch Ophthalmol. 1993 Jan;111(1):104-9. doi: 10.1001/archopht.1993.01090010108035. PMID 7678730
- [Background] Gale CR, Hall NF, Phillips DI, Martyn CN. Lutein and zeaxanthin status and risk of age-related macular degeneration. Invest Ophthalmol Vis Sci. 2003 Jun;44(6):2461-5. doi: 10.1167/iovs.02-0929. PMID 12766044
- [Background] Delcourt C, Carriere I, Delage M, Barberger-Gateau P, Schalch W; POLA Study Group. Plasma lutein and zeaxanthin and other carotenoids as modifiable risk factors for age-related maculopathy and cataract: the POLA Study. Invest Ophthalmol Vis Sci. 2006 Jun;47(6):2329-35. doi: 10.1167/iovs.05-1235. PMID 16723441
- [Background] Tan JS, Wang JJ, Flood V, Rochtchina E, Smith W, Mitchell P. Dietary antioxidants and the long-term incidence of age-related macular degeneration: the Blue Mountains Eye Study. Ophthalmology. 2008 Feb;115(2):334-41. doi: 10.1016/j.ophtha.2007.03.083. Epub 2007 Jul 30. PMID 17664009
- [Background] Cho E, Hankinson SE, Rosner B, Willett WC, Colditz GA. Prospective study of lutein/zeaxanthin intake and risk of age-related macular degeneration. Am J Clin Nutr. 2008 Jun;87(6):1837-43. doi: 10.1093/ajcn/87.6.1837. PMID 18541575
- [Background] VandenLangenberg GM, Mares-Perlman JA, Klein R, Klein BE, Brady WE, Palta M. Associations between antioxidant and zinc intake and the 5-year incidence of early age-related maculopathy in the Beaver Dam Eye Study. Am J Epidemiol. 1998 Jul 15;148(2):204-14. doi: 10.1093/oxfordjournals.aje.a009625. PMID 9676703
- [Background] Cho E, Seddon JM, Rosner B, Willett WC, Hankinson SE. Prospective study of intake of fruits, vegetables, vitamins, and carotenoids and risk of age-related maculopathy. Arch Ophthalmol. 2004 Jun;122(6):883-92. doi: 10.1001/archopht.122.6.883. PMID 15197064
- [Background] Beatty S, Murray IJ, Henson DB, Carden D, Koh H, Boulton ME. Macular pigment and risk for age-related macular degeneration in subjects from a Northern European population. Invest Ophthalmol Vis Sci. 2001 Feb;42(2):439-46. PMID 11157880
- [Background] Bone RA, Landrum JT, Mayne ST, Gomez CM, Tibor SE, Twaroska EE. Macular pigment in donor eyes with and without AMD: a case-control study. Invest Ophthalmol Vis Sci. 2001 Jan;42(1):235-40. PMID 11133874
- [Background] Bernstein PS, Zhao DY, Wintch SW, Ermakov IV, McClane RW, Gellermann W. Resonance Raman measurement of macular carotenoids in normal subjects and in age-related macular degeneration patients. Ophthalmology. 2002 Oct;109(10):1780-7. doi: 10.1016/s0161-6420(02)01173-9. PMID 12359594
- [Background] Obana A, Hiramitsu T, Gohto Y, Ohira A, Mizuno S, Hirano T, Bernstein PS, Fujii H, Iseki K, Tanito M, Hotta Y. Macular carotenoid levels of normal subjects and age-related maculopathy patients in a Japanese population. Ophthalmology. 2008 Jan;115(1):147-57. doi: 10.1016/j.ophtha.2007.02.028. PMID 18166409
- [Background] Hammond BR Jr, Johnson EJ, Russell RM, Krinsky NI, Yeum KJ, Edwards RB, Snodderly DM. Dietary modification of human macular pigment density. Invest Ophthalmol Vis Sci. 1997 Aug;38(9):1795-801. PMID 9286268
- [Background] Berendschot TT, Goldbohm RA, Klopping WA, van de Kraats J, van Norel J, van Norren D. Influence of lutein supplementation on macular pigment, assessed with two objective techniques. Invest Ophthalmol Vis Sci. 2000 Oct;41(11):3322-6. PMID 11006220
- [Background] Bone RA, Landrum JT, Guerra LH, Ruiz CA. Lutein and zeaxanthin dietary supplements raise macular pigment density and serum concentrations of these carotenoids in humans. J Nutr. 2003 Apr;133(4):992-8. doi: 10.1093/jn/133.4.992. PMID 12672909
- [Background] Koh HH, Murray IJ, Nolan D, Carden D, Feather J, Beatty S. Plasma and macular responses to lutein supplement in subjects with and without age-related maculopathy: a pilot study. Exp Eye Res. 2004 Jul;79(1):21-7. doi: 10.1016/j.exer.2004.03.001. PMID 15183097
- [Background] Wenzel AJ, Gerweck C, Barbato D, Nicolosi RJ, Handelman GJ, Curran-Celentano J. A 12-wk egg intervention increases serum zeaxanthin and macular pigment optical density in women. J Nutr. 2006 Oct;136(10):2568-73. doi: 10.1093/jn/136.10.2568. PMID 16988128
- [Background] Bone RA, Landrum JT, Cao Y, Howard AN, Alvarez-Calderon F. Macular pigment response to a supplement containing meso-zeaxanthin, lutein and zeaxanthin. Nutr Metab (Lond). 2007 May 11;4:12. doi: 10.1186/1743-7075-4-12. PMID 17498306
- [Background] Thurnham DI, Tremel A, Howard AN. A supplementation study in human subjects with a combination of meso-zeaxanthin, (3R,3'R)-zeaxanthin and (3R,3'R,6'R)-lutein. Br J Nutr. 2008 Dec;100(6):1307-14. doi: 10.1017/S0007114508971336. Epub 2008 Apr 11. PMID 18405400
- [Background] Huang LL, Coleman HR, Kim J, de Monasterio F, Wong WT, Schleicher RL, Ferris FL 3rd, Chew EY. Oral supplementation of lutein/zeaxanthin and omega-3 long chain polyunsaturated fatty acids in persons aged 60 years or older, with or without AMD. Invest Ophthalmol Vis Sci. 2008 Sep;49(9):3864-9. doi: 10.1167/iovs.07-1420. Epub 2008 Apr 30. PMID 18450596
- [Background] Schalch W, Cohn W, Barker FM, Kopcke W, Mellerio J, Bird AC, Robson AG, Fitzke FF, van Kuijk FJ. Xanthophyll accumulation in the human retina during supplementation with lutein or zeaxanthin - the LUXEA (LUtein Xanthophyll Eye Accumulation) study. Arch Biochem Biophys. 2007 Feb 15;458(2):128-35. doi: 10.1016/j.abb.2006.09.032. Epub 2006 Nov 7. PMID 17084803
- [Background] Trieschmann M, Beatty S, Nolan JM, Hense HW, Heimes B, Austermann U, Fobker M, Pauleikhoff D. Changes in macular pigment optical density and serum concentrations of its constituent carotenoids following supplemental lutein and zeaxanthin: the LUNA study. Exp Eye Res. 2007 Apr;84(4):718-28. doi: 10.1016/j.exer.2006.12.010. Epub 2006 Dec 19. PMID 17306793
- [Background] Johnson EJ, Chung HY, Caldarella SM, Snodderly DM. The influence of supplemental lutein and docosahexaenoic acid on serum, lipoproteins, and macular pigmentation. Am J Clin Nutr. 2008 May;87(5):1521-9. doi: 10.1093/ajcn/87.5.1521. PMID 18469279
- [Background] Zeimer M, Hense HW, Heimes B, Austermann U, Fobker M, Pauleikhoff D. [The macular pigment: short- and intermediate-term changes of macular pigment optical density following supplementation with lutein and zeaxanthin and co-antioxidants. The LUNA Study]. Ophthalmologe. 2009 Jan;106(1):29-36. doi: 10.1007/s00347-008-1773-4. German. PMID 18551295